CLINICAL TRIAL: NCT06950242
Title: Clinical Trial of Safety and Efficacy of Intracranial Laser Balloon Dilation Catheter in Patients With Symptomatic Intracranial Atherosclerotic Stenosis: A Prospective, Multi-center, Randomized Comparison
Acronym: Laser balloon
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (2024) H. 002 (Ss. 01)
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Prospective, Multicenter, Randomized, Controlled, and Superior Efficiency
Keywords: Intracranial Laser Balloon Dilation Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracranial Laser Balloon Dilation Catheter and Laser Generator (Experimental): Experimental group：Name of Medical Apparatus ：Intracranial Laser Balloon Dilation Catheter and Laser Generator Manufacturer：Hangzhou Juzheng Medical Technology limited company
  Interventions: Device: Balloon dilation treatment for intracranial arterial stenosis in order to improve intracranial blood supply.
- Boston Scientific Corporation (Active Comparator): Control group：Name of Medical Apparatus：Gateway PTA Balloon Catheter） Registrant：Boston Scientific Corporation Registration certificate number： CFDA(I) 20193032148
  Interventions: Device: Boston Scientific Corporation

INTERVENTIONS:
Device: Balloon dilation treatment for intracranial arterial stenosis in order to improve intracranial blood supply. — Balloon dilation treatment for intracranial arterial stenosis in order to improve intracranial blood supply.
  Arms: Intracranial Laser Balloon Dilation Catheter and Laser Generator
Device: Boston Scientific Corporation — Balloon dilation treatment for intracranial arterial stenosis in order to improve intracranial blood supply.
  Arms: Boston Scientific Corporation

SUMMARY:
Experimental group：Name of Medical Apparatus ：Intracranial Laser Balloon Dilation Catheter and Laser Generator Manufacturer：Hangzhou Juzheng Medical Technology limited company

DETAILED DESCRIPTION:
This trial is a prospective, multicenter, randomized controlled, high-efficacy clinical trial with a total of 134 participants. Among them, the sample size of randomized controlled trial calculated according to statistics was 128 cases. Patients who require balloon diameter 1.25mm/1.75mm/4.50mm will be assigned to single observation group and treated with intracranial laser balloon dilator catheter combined with laser generator, totaling 6 cases. Subjects who meet the inclusion and exclusion criteria will be randomly assigned to use the intracranial laser balloon dilation catheter produced by Hangzhou Juzheng Medical Technology limited company in combination with a laser generator or the PTA balloon dilation catheter produced by Boston Scientific Company in the control group for the dilation of intracranial arterial stenosis, to verify the effectiveness of the experimental medical device. A clinical summary report will be issued for product registration application after 1-month postoperative follow-up, and a 6-month postoperative follow-up will be conducted to evaluate the medium and long-term efficacy.

The visit nodes for this trial are as follows: screen（Within 15 days before surgery）、 intraoperative、Within 7 days after surgery or before discharge (whichever comes first)、30 days ±7 days after surgery、6 months±30 days after surgery.

This study take immediate postoperative residual stenosis as the primary endpoint to verify the safety and effectiveness of intracranial laser balloon dilator catheter combined with laser generator produced by Hangzhou Juzheng Medical Technology limited company in the treatment of symptomatic intracranial atherosclerotic stenosis patients. The secondary endpoints are the restenosis rate of target lesion, the success rate of surgery, the success rate of instrument, the change of NIHSS score within 7 days after surgery or before discharge, and the change of mRS Score at 6 months after surgery. The incidence of intraoperative device defects, ischemic stroke, hemorrhagic stroke event, mortality, serious adverse events, and adverse events at 30 days and 6 months after surgery were used as safety endpoints to verify the safety and efficacy of the experimental devices.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years old;
2. Symptomatic intracranial artery stenosis, the diameter of the target vessel measured by intracranial angiography was between 70 and 99% (WASID method);
3. The stenosis vessels were in internal carotid artery (intracranial segment), middle cerebral artery, basilar artery, vertebral artery (intracranial segment);
4. The patient had at least one risk factor for intracranial atherosclerosis, including past or existing hypertension, hyperlipidemia, diabetes, smoking, etc.;
5. mRS≤2 before enrollment;
6. 1.25mm≤ target vessel diameter ≤4.5mm;
7. Intracranial artery stenosis requiring interventional treatment was a single lesion;
8. Patients or their guardians can understand the purpose of the trial, voluntarily participate and sign a written informed consent, and can accept follow-up.

Exclusion Criteria:

1. The target vessel is severely calcified and distorted, and the interventional instruments are difficult to be in place or recovered;
2. Acute ischemic stroke occurred within 2 weeks before surgery;
3. Cerebral hemorrhage occurred 3 months before surgery;
4. The target lesion has been treated with interventional therapy before;
5. Intracranial artery stenosis caused by non-atherosclerotic lesions;
6. Intracranial aneurysm or intracranial arteriovenous malformation with an unpredictable high risk or risk of bleeding;
7. Risk factors that may contribute to the risk of cardiogenic embolism (such as left ventricular thrombosis, myocardial infarction within 1 month);
8. History of gastrointestinal bleeding within 6 months;
9. Coagulation dysfunction or obvious bleeding tendency (such as INR > 1.5);
10. Known allergy to contrast agents, anticoagulants, anesthesia and other drugs, red light;
11. Platelet count (PLT<90×109/L);
12. Hemoglobin <100g/L; Uncontrolled severe hypertension (persistent: systolic >180mmHg or diastolic >110mmHg);

(14) Creatinine >3mg/dL, i.e. >265μmol/L; (15) Serious dysfunction of important organs such as heart, liver and kidney; (16) Those who are participating in clinical trials of other drugs or devices that do not meet the primary endpoint; (17) Women who are pregnant or breastfeeding, or who plan to pregnant within one year; (18) Life expectancy is less than 1 year; (19) The researcher determined that there were other circumstances that were not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Immediate residual stenosis after surgery | Time：15 minutes after dilatation of the test or control apparatus.
  Definition：Stenosis of target lesion lumen diameter (%) after test or control instrument dilation (15 minutes).
  Formula： Stenosis of target lesion lumen diameter（%）=（1-Stenosis of target lesion lumen diameter (%) after test or control instrument dilation (15 minutes)）*100%.

SECONDARY OUTCOMES:
Restenosis rate of target lesion after 6 months operation | Time：6 months±30 days after operation
  Definition：DSA examination at 6 months after operation revealed the degree of lumen diameter stenosis of the target lesion>50% and absolute lumen loss>20% of target lesions.
  Formula：degree of diameter stricture（%）=（1-Minimum lumen diameter of target lesion 6 months after surgery/reference vessel diameter of target lesion 6 months after surgery）*100%.
The success rate of operation | Time：15 minutes after dilatation of the test or control apparatus.
  Definition: The proportion of patients with final target lesions with luminal diameter stenosis < 50% and mTICI grade 2b or 3, allowing for the use of additional therapies.
Apparatus success rate | Time：intraoperative
  Definition：The balloon dilatation catheter was successfully delivered in place, the balloon was successfully withdrawn after successful dilatation, the balloon was not ruptured or broken, and there was no equipment failure. The proportion of successful instruments will be calculated.
Changes in NIHSS score within 7 days after surgery or before discharge | 7 days after surgery or before discharge
  The NIHSS score was used to evaluate the functional recovery of the subjects within 7 days after surgery or before discharge.
  Formula：Changes in NIHSS score = NIHSS score within 7 days after surgery or before discharge-baseline NIHSS score。
Changes in mRS at 6 months after surgery | 6 months after operation
  mRS Score was used to evaluate the functional recovery of the subjects at 6 months after operation.
  Formula：Changes in mRS = mRS at 6 months after surgery-baseline mRS score.

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Changzhou., Changzhou, Jiangsu, China